CLINICAL TRIAL: NCT04195594
Title: An Open Label Study to Investigate the Efficacy of Nic's Keto Diet on Cardiovascular Health in Healthy Adults With Mildly Elevated LDL Levels
Brief Title: An Study Investigating Nic's Keto Diet on Cardiovascular Health in Healthy Adults With Mildly Elevated LDL Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TRC GEN+ managed by Trans Russian co Cy (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19KLHT
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Ketogenic Dieting; Healthy
Keywords: Ketogenic Diet; Nic's keto diet; Cardiovascular health; Elevated LDL levels

STUDY DESIGN:
Intervention Model Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nic's Keto Diet (Experimental)
  Interventions: Other: Nic's Keto Diet

INTERVENTIONS:
Other: Nic's Keto Diet — Participants will be instructed to follow Nic's keto diet plan for 140 days. They will be asked to not exceed 20 g of carbohydrates (up to 5% caloric intake) and to consume the remaining 70% of calories from fat sources and 25% from protein sources.

SUMMARY:
The present study will investigate the effects of Nic's Ketogenic diet, comprised of 70% fat, 5% carbohydrate, and 25% protein on middle-aged males and females with mid-range elevated LDL. With the mixed evidence on the causative effect of LDL cholesterol on increased cardiovascular health risk, further studies are warranted to examine the relation of elevated LDL and other biomarkers of cardiovascular health in response to a lifestyle intervention. Furthermore, this study will investigate weight loss and body composition changes with adherence to this dietary intervention over a 140-day period. In this study the efficacy of Nic's Ketogenic diet on weight loss and biomarkers of cardiovascular health will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Provided voluntary, written, informed consent to participate in study
2. Males and females between 30 and 55 years of age
3. BMI between 20.0 to 29.9 kg/m2, inclusive
4. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation) Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. Acceptable methods of birth control include:
   * Non hormonal contraceptives
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
5. Subjects with mid-range (2.5-4.1mmol/L or 100-159 mg/dL) elevated LDL-C levels
6. Agrees to maintain current level of physical activity throughout the study
7. Willingness to complete all questionnaires, records, and diaries and assessments associated with the study and to complete all clinic visits.
8. Healthy as determined by medical history, laboratory results, and as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the course of the trial
2. Women who are menopausal or post-menopausal
3. Currently following a diet (i.e. Ketogenic Diet, low-carbohydrate diet)
4. Subjects with high TSH level (>4.5mU/L) or Self reported pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
5. Participants with type I or II Diabetes Mellitus
6. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable.
7. Participants with previous or current pathology of the pancreas
8. Current or history of Gastroesophageal reflux disease (GERD) or any significant disease of the gastrointestinal tract
9. Self reported hypertension or on hypertensives.
10. Significant cardiovascular event in the past 6 months as assessed by the QI.
11. Major surgery in the past 3 months or individuals who have planned surgery during the course of the trial. Participants with minor surgery will be considered on a case-by-case basis by the QI
12. Gastric bypass surgery
13. Individuals with an autoimmune disease or are immune-compromised
14. Self reported HIV-, Hepatitis B- and/or C-positive diagnosis
15. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones symptom free for 6 months
16. Self reported medical or neuropsychological condition and/or cognitive impairment that, in the QI's opinion, could interfere with study participation
17. Self reported blood/bleeding disorders as per QI
18. Current use of prescribed medications listed in Section 7.3.1
19. Current use of over-the-counter medications, supplements, foods, and/or drinks listed in Section 7.3.2
20. Alcohol or drug abuse within the last 12 months
21. High alcohol intake (>2 standard drinks per day or >10 standard drinks per week)
22. Clinically significant abnormal laboratory results at screening as assessed by the QI
23. Metal implants that may affect the DEXA scan results will be assessed on case-by-case basis by the QI
24. Blood donation 30 days prior to screening, during the study, or a planned donation within 30-days of the last study visit
25. Participation in a clinical research trial within 30 days of study initiation
26. Individuals who are unable to give informed consent
27. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or may pose significant risk to the participant

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

REFERENCES:
- [Derived] Tzenios N, Lewis ED, Crowley DC, Chahine M, Evans M. Examining the Efficacy of a Very-Low-Carbohydrate Ketogenic Diet on Cardiovascular Health in Adults with Mildly Elevated Low-Density Lipoprotein Cholesterol in an Open-Label Pilot Study. Metab Syndr Relat Disord. 2022 Mar;20(2):94-103. doi: 10.1089/met.2021.0042. Epub 2021 Dec 16. PMID 34918971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nic's Keto Diet
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.86 (7.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Eastern European White | 4
  South American | 3
  South Asian | 1
  Western European White | 6
Region of Enrollment [Number; unit: participants]
  Canada | 14

OUTCOME MEASURES:

1. Primary Outcome: Changes to Body Fat Percentage as Assessed by DEXA Scan From Baseline to Day 70 Following Nic's Keto Diet
Description: The DEXA scan is a form of X-ray radiation that measures the body tissue density, which was reported at baseline and compared to day 70.
Time Frame: 70 days
Population: The analysis population takes into account participants that were withdrawn by the qualified investigator and those who were withdrawn at their own request.
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
percentage of body fat | -2.25 (2.48)

2. Primary Outcome: Changes to Muscle Mass Percentage as Assessed by DEXA Scan From Baseline to Day 70 Following Nic's Keto Diet
Description: as for outcome 1
Time Frame: 70 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of muscle mass
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
percentage of muscle mass | 2.24 (2.49)

3. Primary Outcome: Changes to Body Fat Percentage as Assessed by DEXA Scan From Baseline to Day 140 Following Nic's Keto Diet
Description: The DEXA scan is a form of X-ray radiation that measures the body tissue density, which was reported at baseline and compared to day 140.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body fat
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
percentage of body fat | -4.41 (4.04)

4. Primary Outcome: Changes to Muscle Mass Percentage as Assessed by DEXA Scan From Baseline to Day 140 Following Nic's Keto Diet
Description: as for outcome 3
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of muscle mass
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
percentage of muscle mass | 4.38 (4.03)

5. Primary Outcome: Changes to Weight as Assessed by BMI From Baseline to Day 70 Following Nic's Keto Diet
Description: Changes to weight as assessed by BMI was reported at baseline and compared to day 70.
Time Frame: 70 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
kg/m^2 | -1.64 (0.83)

6. Primary Outcome: Changes to Weight as Assessed by BMI From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to weight as assessed by BMI was reported at baseline and compared to day 140.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
kg/m^2 | -2.82 (1.49)

7. Secondary Outcome: The Change in Inflammation, as Assessed by the Change in Erythrocyte Sedimentation Rate (ESR) Following Nic's Keto Diet for 140 Days
Description: The change in inflammation, as assessed by the change in erythrocyte sedimentation rate (ESR) following Nic's Keto Diet was reported at 140 days.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mm/hr | 0.36 (4.43)

8. Secondary Outcome: The Change in Inflammation, as Assessed by the Change in C-reactive Protein (CRP) Following Nic's Keto Diet for 140 Days
Description: The change in inflammation, as assessed by the change in C-reactive protein (CRP) following Nic's Keto Diet was reported at 140 days.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mg/L | -0.71 (2.10)

9. Secondary Outcome: Changes to Weight From Baseline to Day 28 Following Nic's Keto Diet
Description: Changes to weight from baseline were reported and compared to day 28 following Nic's Keto Diet.
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
kg | -3.02 (2.09)

10. Secondary Outcome: Changes to Weight From Baseline to Day 56 Following Nic's Keto Diet
Description: Changes to weight from baseline were reported and compared to day 56 following Nic's Keto Diet.
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
kg | -4.47 (2.79)

11. Secondary Outcome: Changes to Weight From Baseline to Day 84 Following Nic's Keto Diet
Description: Changes to weight from baseline were reported and compared to day 84 following Nic's Keto Diet.
Time Frame: 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
kg | -5.58 (3.07)

12. Secondary Outcome: Changes to Weight From Baseline to Day 112 Following Nic's Keto Diet
Description: Changes to weight from baseline were reported and compared to day 112 following Nic's Keto Diet.
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
kg | -6.43 (3.93)

13. Secondary Outcome: Changes to Systolic Blood Pressure From Baseline to Day 28 Following Nic's Keto Diet
Description: Changes to systolic blood pressure from baseline were reported and compared to day 28 following Nic's Keto Diet.
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mm Hg | 1.23 (7.79)

14. Secondary Outcome: Changes to Systolic Blood Pressure From Baseline to Day 56 Following Nic's Keto Diet
Description: Changes to systolic blood pressure from baseline were reported and compared to day 56 following Nic's Keto Diet.
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mm Hg | -3.06 (6.62)

15. Secondary Outcome: Changes to Systolic Blood Pressure From Baseline to Day 84 Following Nic's Keto Diet
Description: Changes to systolic blood pressure from baseline were reported and compared to day 84 following Nic's Keto Diet.
Time Frame: 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mm Hg | -2.73 (8.30)

16. Secondary Outcome: Changes to Systolic Blood Pressure From Baseline to Day 112 Following Nic's Keto Diet
Description: Changes to systolic blood pressure from baseline were reported and compared to day 112 following Nic's Keto Diet.
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mm Hg | -3.85 (7.58)

17. Secondary Outcome: Changes to Systolic Blood Pressure From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to systolic blood pressure from baseline were reported and compared to day 140 following Nic's Keto Diet.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mm Hg | -6.52 (9.53)

18. Secondary Outcome: Changes to Total Cholesterol From Baseline to Day 28 Following Nic's Keto Diet
Description: Changes to total cholesterol were reported from baseline and compared to day 28 following Nic's Keto diet using blood analysis (units in mmol/L)
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.87 (1.01)

19. Secondary Outcome: Changes to Triglyceride Level From Baseline to Day 28 Following Nic's Keto Diet
Description: Changes to triglyceride level were reported from baseline and compared to day 28 following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.04 (0.62)

20. Secondary Outcome: Changes to HDL-Cholesterol From Baseline to Day 28 Following Nic's Keto Diet
Description: Changes to HDL-cholesterol from baseline to day 28 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | -0.04 (0.27)

21. Secondary Outcome: Changes to LDL-Cholesterol From Baseline to Day 28 Following Nic's Keto Diet
Description: Changes to LDL-cholesterol from baseline to day 28 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.89 (0.84)

22. Secondary Outcome: Changes to Total Cholesterol From Baseline to Day 56 Following Nic's Keto Diet
Description: Changes to total cholesterol from baseline to day 56 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.91 (0.97)

23. Secondary Outcome: Changes to Triglyceride Level From Baseline to Day 56 Following Nic's Keto Diet
Description: Changes to triglyceride level from baseline to day 56 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | -0.07 (0.67)

24. Secondary Outcome: Changes to HDL-Cholesterol From Baseline to Day 56 Following Nic's Keto Diet
Description: Changes to HDL-Cholesterol from baseline to day 56 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.01 (0.28)

25. Secondary Outcome: Changes to LDL-Cholesterol From Baseline to Day 56 Following Nic's Keto Diet
Description: Changes to LDL-Cholesterol from baseline to day 56 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.93 (0.87)

26. Secondary Outcome: Changes to Total Cholesterol From Baseline to Day 84 Following Nic's Keto Diet
Description: Changes to total cholesterol from baseline to day 84 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mmol/L | 1.13 (1.21)

27. Secondary Outcome: Changes to Triglyceride Level From Baseline to Day 84 Following Nic's Keto Diet
Description: Changes to triglyceride level from baseline to day 84 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mmol/L | -0.11 (0.57)

28. Secondary Outcome: Changes to HDL-Cholesterol From Baseline to Day 84 Following Nic's Keto Diet
Description: Changes to HDL-Cholesterol from baseline to day 84 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mmol/L | 0.02 (0.32)

29. Secondary Outcome: Changes to LDL-Cholesterol From Baseline to Day 84 Following Nic's Keto Diet
Description: Changes to LDL-Cholesterol from baseline to day 84 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mmol/L | 1.16 (1.12)

30. Secondary Outcome: Changes to Total Cholesterol From Baseline to Day 112 Following Nic's Keto Diet
Description: Changes to total cholesterol from baseline to day 112 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | 1.01 (1.31)

31. Secondary Outcome: Changes to Triglyceride Level From Baseline to Day 112 Following Nic's Keto Diet
Description: Changes to triglyceride level from baseline to day 112 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | -0.16 (0.55)

32. Secondary Outcome: Changes to HDL-Cholesterol From Baseline to Day 112 Following Nic's Keto Diet
Description: Changes to HDL-Cholesterol from baseline to day 112 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | 0.10 (0.38)

33. Secondary Outcome: Changes to LDL-Cholesterol From Baseline to Day 112 Following Nic's Keto Diet
Description: Changes to LDL-Cholesterol from baseline to day 112 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | 0.99 (1.17)

34. Secondary Outcome: Changes to Total Cholesterol From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to total cholesterol from baseline to day 140 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | 1.06 (1.10)

35. Secondary Outcome: Changes to Triglyceride Level From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to triglyceride level from baseline to day 140 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | -0.23 (0.41)

36. Secondary Outcome: Changes to HDL-Cholesterol From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to HDL-Cholesterol from baseline to day 140 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | 0.15 (0.27)

37. Secondary Outcome: Changes to LDL-Cholesterol From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to LDL-Cholesterol from baseline to day 140 were reported following Nic's Keto diet using blood analysis (units in mmol/L).
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | 1.02 (0.94)

38. Secondary Outcome: Changes to HbA1c From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to HbA1c were reported at baseline and compared to day 140 following Nic's Keto Diet.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of Glycosylated Haemoglobin
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
percent of Glycosylated Haemoglobin | -0.22 (0.18)

39. Secondary Outcome: Changes to Fasting Glucose From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to fasting glucose were reported at baseline and compared to day 140 following Nic's Keto Diet.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mmol/L | -0.06 (0.37)

40. Secondary Outcome: Changes to Free Tri-iodothyronine (T3) From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to free tri-iodothyronine (T3) were reported at baseline and compared to day 140 following Nic's Keto Diet.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
pmol/L | -0.85 (0.55)

41. Secondary Outcome: Changes to Weight From Baseline to Day 70 Following Nic's Keto Diet
Description: Changes to weight were reported from baseline and compared to day 70 following Nic's Keto Diet.
Time Frame: 70 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
kg | -4.90 (2.66)

42. Secondary Outcome: Changes to Weight From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to weight were reported from baseline and compared to Day 140 following Nic's Keto Diet.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
kg | -8.55 (4.74)

43. Secondary Outcome: Changes to Systolic Blood Pressure From Baseline to Day 70 Following Nic's Keto Diet
Description: Changes to systolic blood pressure were reported from baseline and compared to Day 70 following Nic's Keto Diet.
Time Frame: 70 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mm Hg | -3.72 (7.96)

44. Secondary Outcome: Changes to Diastolic Blood Pressure From Baseline to Day 28 Following Nic's Keto Diet
Description: Changes to diastolic blood pressure were reported from baseline and compared to Day 28 following Nic's Keto Diet.
Time Frame: 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mm Hg | 3.23 (6.06)

45. Secondary Outcome: Changes to Diastolic Blood Pressure From Baseline to Day 56 Following Nic's Keto Diet
Description: Changes to diastolic blood pressure were reported from baseline and compared to Day 56 following Nic's Keto Diet.
Time Frame: 56 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mm Hg | 0.44 (5.13)

46. Secondary Outcome: Changes to Diastolic Blood Pressure From Baseline to Day 70 Following Nic's Keto Diet
Description: Changes to diastolic blood pressure were reported from baseline and compared to Day 70 following Nic's Keto Diet.
Time Frame: 70 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 12
mm Hg | -0.14 (6.81)

47. Secondary Outcome: Changes to Diastolic Blood Pressure From Baseline to Day 84 Following Nic's Keto Diet
Description: Changes to diastolic blood pressure were reported from baseline and compared to Day 84 following Nic's Keto Diet.
Time Frame: 84 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mm Hg | -2.33 (7.34)

48. Secondary Outcome: Changes to Diastolic Blood Pressure From Baseline to Day 112 Following Nic's Keto Diet
Description: Changes to diastolic blood pressure were reported from baseline and compared to Day 112 following Nic's Keto Diet.
Time Frame: 112 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mm Hg | -1.21 (5.25)

49. Secondary Outcome: Changes to Diastolic Blood Pressure From Baseline to Day 140 Following Nic's Keto Diet
Description: Changes to diastolic blood pressure were reported from baseline and compared to Day 140 following Nic's Keto Diet.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
mm Hg | 0.30 (6.60)

50. Other Pre Specified Outcome: Number of Pre-emergent and Post-emergent Adverse Events
Description: Number of pre-emergent and post-emergent adverse events (AEs)
Time Frame: 140 days
Population: Safety population
Measure: Number; unit: events
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 14
events | 44

51. Other Pre Specified Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Readings After 70 Days Following Nic's Keto Diet
Description: ECG reports will be analysed after 70 days of following Nic's Keto Diet and compared to baseline. All ECGs will be assessed by the Qualified Investigator on a case-by-case basis to determine if they were normal or abnormal based on the full clinical picture and patient details. Number of participants with clinically relevant abnormal ECGs will be recorded.
Time Frame: 70 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 14
participants | 0

52. Other Pre Specified Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Readings After 140 Days Following Nic's Keto Diet
Description: ECG reports will be analysed after 140 days of following Nic's Keto Diet and compared to baseline. All ECGs will be assessed by the Qualified Investigator on a case-by-case basis to determine if they were normal or abnormal based on the full clinical picture and patient details. Number of participants with clinically relevant abnormal ECGs will be recorded.
Time Frame: 140 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 14
participants | 0

53. Other Pre Specified Outcome: Change in Heart Rate After 140 Days of Following Nic's Keto Diet
Description: Changes in heart rate after 140 days of following Nic's Keto Diet and compared to baseline.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
bpm | 0.61 (9.06)

54. Other Pre Specified Outcome: Change in Body Mass Index (BMI) After 140 Days of Following Nic's Keto Diet
Description: Change in Body Mass Index (BMI) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 11
kg/m^2 | -2.82 (1.49)

55. Other Pre Specified Outcome: Change in Alanine Aminotransferase (ALT) After 140 Days of Following Nic's Keto Diet
Description: Change in alanine aminotransferase (ALT) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: The analysis population takes into account participants that were withdrawn by the qualified investigator and/or those who were withdrawn at their own request.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
U/L | -1.01 (7.82)

56. Other Pre Specified Outcome: Change in Aspartate Aminotransferase (AST) After 140 Days of Following Nic's Keto Diet
Description: Change in aspartate aminotransferase (AST) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
U/L | 0.08 (6.95)

57. Other Pre Specified Outcome: Change in Total Bilirubin After 140 Days of Following Nic's Keto Diet
Description: Change in total bilirubin after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
µmol/L | 0.23 (5.63)

58. Other Pre Specified Outcome: Change in Creatinine After 140 Days of Following Nic's Keto Diet
Description: Change in creatinine after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
µmol/L | 3.77 (9.58)

59. Other Pre Specified Outcome: Change in Sodium Electrolyte Levels After 140 Days of Following Nic's Keto Diet
Description: Change in sodium electrolyte levels after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.92 (2.33)

60. Other Pre Specified Outcome: Change in Potassium Electrolyte Levels After 140 Days of Following Nic's Keto Diet
Description: Change in potassium electrolyte levels after 140 days of following Nic's Keto Diet
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | -0.12 (0.46)

61. Other Pre Specified Outcome: Change in Chloride Electrolyte Levels After 140 Days of Following Nic's Keto Diet
Description: Change in chloride electrolyte levels after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | -0.23 (1.92)

62. Other Pre Specified Outcome: Change in Phosphorus Electrolyte Levels After 140 Days of Following Nic's Keto Diet
Description: Change in phosphorus electrolyte levels after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mmol/L | 0.14 (0.16)

63. Other Pre Specified Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) After 140 Days of Following Nic's Keto Diet
Description: Change in estimated glomerular filtration rate (eGFR) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
mL/min/1.73m^2 | -5.00 (11.08)

64. Other Pre Specified Outcome: Change in Amount of Neutrophils After 140 Days of Following Nic's Keto Diet
Description: Change in amount of neutrophils after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: x10^9 neutrophils/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
x10^9 neutrophils/L | -0.53 (1.21)

65. Other Pre Specified Outcome: Change in Amount of Lymphocytes After 140 Days of Following Nic's Keto Diet
Description: Change in amount of lymphocytes after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: x10^9 lymphocytes/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
x10^9 lymphocytes/L | -0.17 (0.47)

66. Other Pre Specified Outcome: Change in Amount of Monocytes After 140 Days of Following Nic's Keto Diet
Description: Change in amount of monocytes after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: x10^9 monocytes/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
x10^9 monocytes/L | -0.06 (0.14)

67. Other Pre Specified Outcome: Change in Amount of Eosinophils After 140 Days of Following Nic's Keto Diet
Description: Change in amount of eosinophils after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: x10^9 eosinophils/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
x10^9 eosinophils/L | 0.00 (0.08)

68. Other Pre Specified Outcome: Change in Amount of Basophils After 140 Days of Following Nic's Keto Diet
Description: Change in amount of basophils after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: x10^9 basophils/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
x10^9 basophils/L | 0.00 (0.04)

69. Other Pre Specified Outcome: Change in Red Blood Cell (RBC) Count After 140 Days of Following Nic's Keto Diet
Description: Change in red blood cell (RBC) count after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: x10^12 RBC/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
x10^12 RBC/L | -0.05 (0.20)

70. Other Pre Specified Outcome: Change in Hemoglobin Levels After 140 Days of Following Nic's Keto Diet
Description: Change in hemoglobin levels after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
g/L | -1.46 (6.31)

71. Other Pre Specified Outcome: Change in Hematocrit Levels After 140 Days of Following Nic's Keto Diet
Description: Change in hematocrit levels after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: l/l
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
l/l | 0.00 (0.02)

72. Other Pre Specified Outcome: Change in Platelet Count After 140 Days of Following Nic's Keto Diet
Description: Change in platelet count after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: x10^9 platelets/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
x10^9 platelets/L | 15.85 (30.56)

73. Other Pre Specified Outcome: Change in Mean Corpuscular Volume (MCV) After 140 Days of Following Nic's Keto Diet
Description: Change in mean corpuscular volume (MCV) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: fl
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
fl | 0.85 (1.41)

74. Other Pre Specified Outcome: Change in Mean Corpuscular Hemoglobin (MCH) After 140 Days of Following Nic's Keto Diet
Description: Change in mean corpuscular hemoglobin (MCH) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
pg | -0.08 (0.95)

75. Other Pre Specified Outcome: Change in Mean Corpuscular Hemoglobin Concentration (MCHC) After 140 Days of Following Nic's Keto Diet
Description: Change in mean corpuscular hemoglobin concentration (MCHC) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
g/L | -3.69 (7.48)

76. Other Pre Specified Outcome: Change in Red Cell Distribution Width (RDW) After 140 Days of Following Nic's Keto Diet
Description: Change in red cell distribution width (RDW) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: percentage of variation
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
percentage of variation | 0.37 (0.71)

77. Other Pre Specified Outcome: Change in Mean Platelet Volume (MPV) After 140 Days of Following Nic's Keto Diet
Description: Change in mean platelet volume (MPV) after 140 days of following Nic's Keto Diet compared to baseline.
Time Frame: 140 days
Population: as for outcome 55
Measure: Mean (Standard Deviation); unit: fl
Arm/Group | Nic's Keto Diet
Number analyzed (Participants) | 13
fl | -0.20 (0.26)

ADVERSE EVENTS:
Time Frame: 140 days
Description: During the study, participants recorded AEs in their diary. At each visit, the participant was asked "have you experienced any difficulties or problems since I last saw you?" upon which answers (AEs) were documented in the study record and were classified as per the description, duration, intensity, frequency, and outcome. The qualified investigator assessed any AEs and decided causality.
Arm/Group | Nic's Keto Diet
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nic's Keto Diet (N=14)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Amenorrhoea (Endocrine disorders) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Sleep disorder (Psychiatric disorders) | 4 (4)
Insomnia (Nervous system disorders) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Oropharyngeal pain (Gastrointestinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Vessel puncture site bruise (Vascular disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is an employee of the CRO that conducted the study. The research agreement indicates that the data is the property of the sponsor and therefore they control the option for disclosing results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04195594/Prot_SAP_000.pdf